CLINICAL TRIAL: NCT03457064
Title: Enhancing Physical Activity With a Social Support Adherence Intervention
Brief Title: Physical Activity With Social Support Adherence Intervention
Acronym: PASAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Jiska Cohen-Mansfield (Other)
Responsible Party: Sponsor-Investigator, Professor Jiska Cohen-Mansfield, Professor, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TelAvivUniv
Record Dates: First submitted 2018-02-20; First posted 2018-03-07 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Sedentary Status of Older Adults
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (PA) (No Intervention): Physical activity (PA) involved a program of physical exercise alone.
- PA+Social Adherence Intervention(PASAI) (Active Comparator): PA+Social Adherence Intervention(PASAI) involved a program of physical exercise combined with a social adherence intervention.
  Interventions: Behavioral: PA+Social Adherence Intervention(PASAI)

INTERVENTIONS:
Behavioral: PA+Social Adherence Intervention(PASAI) — While both physical activity programs were tailored to match participants' physical needs and abilities, the PA+Social Adherence Intervention(PASAI) introduced elements to promote and strengthen self-efficacy and social interaction among participants.
  Other Names: Physical Activity (PA)
  Arms: PA+Social Adherence Intervention(PASAI)

SUMMARY:
The study compares two programs to increase physical activity among sedentary old persons. The first is a provision of a free physical activity program tailored to their abilities. The other combines the same free physical activity with an adherence intervention which focuses on social contact with others in the program and on enhancing self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary older adults.
* Residents in congregate housing.

Exclusion Criteria:

* Age under 70.
* Not completing an informed consent form.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the Rapid Assessment of Physical Activity (RAPA). | Baseline and Three Months.
  RAPA is an easily administered nine item questionnaire developed to assess physical activity levels among older adults.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen-Mansfield J, Sommerstein M. Motivating Inactive Seniors to Participate in Physical Activity: A Pilot RCT. Am J Health Behav. 2019 Jan 1;43(1):195-206. doi: 10.5993/AJHB.43.1.16. PMID 30522577